CLINICAL TRIAL: NCT00168168
Title: ACB A Randomized Study of 2.5ug/kg/Day vs. 5ug/kg/Day Dose of G-CSF After High Dose Chemotherapy Followed by Autologous Peripheral Blood Stem Cell/Marrow Transplant Recipients FILE#17159
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HE-10-0053
Record Dates: First submitted 2005-09-14; First posted 2005-09-15 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2007-04

CONDITIONS: Peripheral Stem Cell/Marrow Transplant
Keywords: G-CSF; Filgrastim; Engraftment time; Autologus transplant

INTERVENTIONS:
Drug: G-CSF/Filgrastim

SUMMARY:
Evaluate recovery time on 2.5 mg/Kg/day dose of G-CSF versus 5 mg/Kg/day dose.

ELIGIBILITY:
Inclusion Criteria:

* over age 18
* autologous stem cell/marrow transplant candidate in MM, lymphoma, AMG and testicular

Exclusion Criteria:

* age below 18 years
* sensitive to G-CSF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-07; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meluka Game, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada